CLINICAL TRIAL: NCT04317755
Title: A Randomised Control Trial Evaluating a Comic-based School Intervention to Promote Body Confidence and Related Outcomes Among Adolescents in India
Brief Title: Evaluation of the Impact of a Comic-based Programme to Promote Body Confidence Among Adolescents in India
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the West of England (Other)
Collaborators: Unilever R&D (Industry); UNICEF (Other); BBC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HAS-HSS-18-098
Record Dates: First submitted 2020-02-05; First posted 2020-03-23 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Body Image; Eating Disorder Symptom

STUDY DESIGN:
Intervention Model Description: Parallel 2-arm cluster randomised controlled trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Masking not possible for participants within design, but investigators and outcome assessors will not know what condition participants are assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Comic-based body image programme
  Interventions: Behavioral: AdhaFULL body image comics
- Control (No Intervention): Schools lessons as usual

INTERVENTIONS:
Behavioral: AdhaFULL body image comics — The comics were co-created with the expertise of four stakeholders: the investigators, UNICEF, BBC Media Action, and the Dove Self-Esteem Project. There are six different comics, which target issues relating to gender stereotypes and appearance concerns amongst adolescents in rural India. Based on 'Dove Confident Me', each comic tells a story which targets a specific established risk factor for body dissatisfaction. Specifically, they focus on gender prejudice (Comic 1), societal appearance ideals (Comic 2), media literacy (Comic 3), appearance comparisons (Comic 4), appearance-related conversations and teasing (Comic 5), and promoting 'body activism' (Comic 6). In each session, students will read the respective comic as a class. At the end of each comic, the teacher will facilitate one or two activities with the students based on the key learnings from the comics. These activities will encourage students to think critically about what they have read and consolidate their learning.
  Arms: Intervention

SUMMARY:
Body dissatisfaction is a leading concern for young people and can have serious health consequences. Emerging approaches for improving body image are effective among adolescents in the school setting. However, the majority of trials are conducted in high-income westernised countries, despite body dissatisfaction being increasingly recognised as a global concern. As such, it is important to develop and disseminate interventions to promote body confidence among adolescents in in low-to-middle income countries, too.

One country where body image concerns are becoming an increasing issue is India. The investigators recently finished developing and evaluating a body image programme among adolescents in New Delhi, India; which found immediate and 3-month improvements in body image, disordered eating, self-esteem, and other related outcomes. Whilst these findings offer an effective body image programme for school students in urban areas of India, this may not be feasible for schools in more rural and lower socio-economic areas in India.

The aim of the present study is therefore to conduct an acceptability study, followed by a randomised controlled trial (RCT), of a comics-based body image programme among adolescents in a semi-rural area of India (Rajasthan), in order to understand its acceptability, feasibility, and preliminary efficacy. This comic-based programme will be based on Dove Confident Me, which was found to be effective among adolescents in Delhi, India.

To assess the acceptability of the comic-book-based programme, interviews and focus groups will be conducted with students and teachers. This in-depth feedback will be used to optimise the programme. Next, an RCT will compare body image and well-being of students who take part in the programme to students who do not take part (classes as usual) to examine the programme's efficacy. The investigators will recruit students and teachers from schools in a rural and lower socio-economic area of India (Rajasthan). Students will complete questionnaire assessments of body image and well-being before and after the 6-session intervention (across 4 weeks), and again at 3-month follow-up to assess longer-term benefits.

It is hypothesised that students who receive the intervention will have better body image and wellbeing relative to the control group at both post-intervention and follow-up.

DETAILED DESCRIPTION:
Background:

Body image is a significant and prevalent concern for adolescents in high-income countries such as the UK, the USA, and Australia. For example, a national survey of nearly 22,000 young people in Australia found that 3 in 10 adolescent boys and girls are concerned about their appearance. This high prevalence of body image concerns is worrisome, given their serious negative physical and psychological health consequences, including unhealthy weight loss behaviours, eating disorders, depression and self-harm, substance use, and lower levels of academic engagement.

There is increasing recognition that body dissatisfaction is a global issue. For example, in India, 57% of adolescents report being concerned with their appearance. Further, girls across different regions of India have expressed concerns in relation to their weight and report dieting behaviours. Skin colour has also been indicated as an additional source of appearance concern among young people in India. Indeed, research indicated that 19% of Indian undergraduate students had used a skin lightening product in the previous 12 months, strongly suggesting dissatisfaction with their natural skin tone, which may be pertinent to younger groups.

Collectively, these findings indicate the importance of developing and disseminating interventions to promote positive body image among adolescents in India. The investigators recently finished developing and evaluating a school-based body image programme, 'Dove Confident Me', among adolescents in New Delhi, India. Immediate and 3-month follow-up improvements were found in body image, disordered eating, self-esteem, and other related outcomes. Whilst these findings offer an effective body image programme for school students in urban areas of India, this may not be feasible for schools in more rural and lower socio-economic areas in India, where there is limited electricity and computers.

Therefore, the aim of the present study is to conduct an acceptability study followed by a randomised controlled trial of a comic-based body image programme among adolescents in a semi-rural area of India (Rajasthan), in order to understand its acceptability, feasibility, and preliminary efficacy. This comic-book-based programme will be based on 'Dove Confident Me'.

It is hypothesised that students who receive the comic-based body image intervention will experience immediate and sustained improvements in the primary (i.e., body image) and secondary outcomes (i.e., eating pathology, internalisation of appearance ideals, body image-related life disengagement, self-esteem, positive and negative mood) relative to students in the control condition. There are no hypotheses in relation to the impact of the intervention on the exploratory outcomes (I.e., skin colour dissatisfaction, body hair dissatisfaction, appearance-based teasing, endorsement of traditional gender norms).

Study 1: Acceptability study

Study design

A qualitative approach will be adopted to explore students' and teachers' acceptability (i.e., thoughts and feedback) on the comics. Online interviews will be conducted with students, whilst online focus groups will be conducted with teachers, both informed by a semi-structured interview schedule. All participants will also be asked a series of quantitative questions exploring acceptability of the comics.

Recruitment and participants

The Department of Education in Rajasthan will select one school which meets the inclusion criteria to participate in the research (see elsewhere). A total of nine teachers who teach across Classes 6-8 (three teachers from each year group) will be invited to participate in an online focus group (five teachers in one focus group, four teachers in a second focus group). However, a total of 36 students across Classes 6-8 (aged 11-14 years) will be invited to participate in online interviews, whereby the first nine interviews will help in theme identification and the remaining 27 interviews will contribute towards developing a greater understanding of each theme. This sample will be equally divided across the three years, genders, and reading and writing proficiency, which will be assessed by their teachers. This will lead to six girls and six boys in each year group, with three boys and three girls with a higher level of reading and writing proficiency, and three boys and three girls with a lower level of reading and writing proficiency.

Procedure

On behalf of the authors, who are unable to travel to India due to the COVID-19 pandemic, an International Organization for Standardisation-(ISO)-certified research agency will collect data. Once parents have provided consent for their children to participate in the study, students will provide informed assent. Teachers will be provided with information about the study and a consent form. Next, each participant will be sent a copy of the six comics to read at home. A week later, the research agency will conduct the online focus groups with teachers and online interviews with students. The interviews and focus groups will be audio-recorded and last between 45-60 minutes. Participants will then be asked to complete the brief quantitative questionnaire.

Data analysis

A Data Management Plan will be prepared in line with requirements of university research governance. Audio-recordings will be transcribed verbatim and anonymized. Transcripts will be simultaneously analysed by two of the authors using qualitative codebook thematic analysis. Questionnaire data will be entered into an SPSS file, and descriptive analyses will be conducted on the data. Findings from both the qualitative and quantitative data will be used to optimise the comics and Teacher Guides prior to their evaluation in the randomised controlled trial (RCT).

Study 2: RCT

Trial design

A parallel two-arm, cluster RCT will be employed to evaluate the AdhaFULL comic-based intervention. Schools will be randomized before completion of T1 data collection. The study design comprises two independent groups with outcome data collected at three time points (T1, T2, T3). T1 is baseline (Week 1); T2 is 1-week post-intervention (Week 5) at the end of intervention; T3 is 12-weeks follow-up (Week 16). The resulting data is amenable to standard analysis for two group comparisons including a 2 by 2 by 2 by mixed factorial design with randomized group as a two level between subjects fixed factor, trial phase (T2, T3) as a longitudinal two-level repeated measures factor, gender as a two-level fixed factor and with the commensurate baseline measure (T1) as a mean adjusted covariate. Randomized school will be a random factor in the analyses. Following T3 data collection, schools in the control condition will receive all intervention materials, including the training documents for teachers.

Recruitment and participants

Government schools in Rajasthan will be recruited using stratified sampling based on two key sociodemographic factors: the degree of ruralness of the area within which the school is located, the school's exam results. The main recruitment sites will be identified by Rajasthan's Department of Education, who will select schools that meet the inclusion criteria (see elsewhere). Once the school principal provides consent to participate in the research, each school will be randomly allocated to either the intervention or lessons-as-usual control condition. Students in Classes 6-8 (aged 11 to 14 years) will be invited to participate in the study.

Sample size calculations

The evaluation of 'Dove Confident Me' in an urban Indian setting indicated a range of effect sizes for outcome measures with standardized effects in the small to medium range and exceeding an effect size of d = 0.2, which would minimally be of interest to public health policy makers (Lewis-Smith et al., Under review). For a lower bound of d = 0.2, a sample size of n = 540 boys and n = 540 girls per arm would have 95% power to detect an effect separately for each gender (two-sided, alpha = 0.05). To account for 10% loss, the sample size will be inflated by (540/10 =) 54 of each gender per arm, and to account for 10% loss within this additional recruitment, a further inflation of (54/10 =) 6 to give a target sample size of 600 boys and 600 girls per arm, totalling 1,200 per arm (intervention versus control). Therefore, a total of 2,400 students will be recruited. Students will be equally divided across years 6,7, and 8, and gender.

Randomization

Participants will be randomized to either the intervention or control arm at the school level. Randomization will be conducted at the school level to avoid spill over effects due to communication about the intervention to the control group. Eligible schools will be randomised in a target 1:1 ratio using minimization with a residual error. The minimization factors are (i) number of students at grade 6, 7 or 8 and (ii) proportion of boys at grade 6, 7, and 8. The first 8 schools will be allocated using blocked randomisation thereafter probabilistic minimization will occur with the probability of minimizing set to 0.8.

Outcome measures

There are very few body image and related psychological outcome measures which have undergone rigorous validation in India, and those which have, tend to be in English. The outcome measures that will be used in this trial are currently being validated in Hindi by the investigators, with rigorous steps employed (Swami & Barron, 2019). The validation will be completed prior to commencing the present study. Thus, the final items may differ from those in the original scales below and will be reported in the main trial paper (see outcome measures elsewhere).

Since the original protocol, concerns regarding the sample's ability to comprehend the measures led to the addition of more visual and less literacy-dependent exploratory measures, which are described under the 'Outcome Measures' section.

Other measures

Demographics

Demographic information will be collected from students in the T1 questionnaire, including age, gender, religion, language spoken at home, the family's primary wage earner's level of education, parents' occupations, number of bedrooms in the house, and whether certain electronic items are owned by the household (e.g., television, computer). The socio-economic status of participants will be estimated using India's New Consumer Classification System (NCCS; Kakati & Ahmed, 2016).

Intervention acceptability

Acceptability of the comic-based intervention will again be assessed among students in the intervention condition via the T2 questionnaire. They will be asked to indicate their degree of agreement or disagreement using a five-point Likert scale (1 = Strongly disagree to 5 = Strongly agree) with statements concerning their perceptions of the intervention (e.g., "I enjoyed the lessons", "I understood what was being taught in the lessons", "I think adolescents would find the activities beneficial and interesting"). Teachers will also be asked to complete a brief questionnaire to assess intervention acceptability. They will be asked to indicate their degree of agreement or disagreement using a five-point Likert scale (1 = Strongly disagree to 5 = Strongly agree) with statements regarding their perceptions of intervention delivery and student engagement (e.g., "I enjoyed delivering these lessons", "Students understood the key messages of these lessons", "I felt confident delivering these sessions"). A subgroup of teachers and students will be invited to participate in separate focus groups or interviews, to explore intervention acceptability in greater depth from both perspectives.

Attention checks

To assess the degree of attention from participants whilst completing each questionnaire, attention checks will be embedded throughout at all three time-points. These items will instruct participants to select a specific response on a Likert scale (e.g., Please select 'Strongly Agree'). There will also be attention checks which are specific to each comic's storyline in the T2 survey. These will be used to assess participants' recall of the comics and to determine the number of participants that were present in each session. There will be a question about each comic (e.g., "Why does Seema's mother stop her from playing outside?"), to which participants will need to select the correct answer from four options (e.g., "she wants Seema to study for school", "she says it's too dark to play outside", "I did not attend Session 1/do not recognize the story").

Intervention fidelity A proportion of sessions will be observed by researchers, and teachers will be asked to audio-record the delivery of their sessions. Fidelity assessment will be based on previous school intervention evaluation studies (Garbett et al., 2021; Diedrichs et al., 2021), whereby a standardised checklist will assess three domains: perceived facilitator competence, the extent to which learning outcomes were met, and adherence to the intervention. Sessions with both audio and live observation will be used to assess interrater reliability.

Procedure

Ethical guidelines for conducting anonymous public health research in India (Indian Council of Medical Research, 2018) indicate that parental consent is sought at the school's discretion. However, with the permission of Department of Education of Rajasthan in India, parents will be given two weeks to provide opt-out consent. Additionally, the children will be provided with information about the study and given the opportunity to ask questions before they indicate written assent. The research agency will liaise with each recruited school to decide on an alternative activity for the students without consent/assent. This will take place outside of the classroom where the intervention is being delivered or data collection is occurring. Once all consent procedures have been completed, a team of trained researchers from an ISO-certified research agency will administer T1 outcome assessments via a self-report paper survey with all students irrespective of randomized arm. All students will complete the surveys in a quiet classroom in the presence of a researcher and schoolteacher and will be encouraged to complete the questions independently (T1). Further outcome assessments will be administered via paper questionnaires in the week following the final session of the intervention (T2) and at 12-weeks follow-up (T3). Once outcome assessments have been completed by students, the data will be entered into a password-protected Excel spreadsheet, and subsequently imported into an SPSS data file for analysis. A Data Management Plan will be prepared in line with requirements of university research governance. This data will be stored on a secure encrypted network on the university system.

With regard to intervention delivery, a 'train-the-trainer' approach will be adopted. This will involve having expert trainers (i.e, the authors, who are experienced in the train-the-trainer approach) teach non-expert providers (i.e., the research agency) how to subsequently train teachers in delivery of the intervention. The train-the-teacher approach has demonstrated efficacy in previous body image intervention evaluations and facilitates scalability and sustainability. The research agency will receive a two-day training course, and subsequently, teachers will receive a one-day training course. The teacher training will cover the theoretical basis of the intervention, including risk factors for body dissatisfaction, and the associated consequences. Subsequently, the teachers will be familiarised with the comics and associated activities and will participate in role plays to practise delivering the intervention. Finally, they will be given hints and tips for delivering the sessions and practise answering challenging questions that could be posed by the students. All schools in the intervention condition will begin the intervention in the week following T1 outcome assessment. Teachers will deliver each session during a school lesson, and the six sessions will be delivered at a rate of two sessions per week. Each session will begin with the teacher reading the comic with the class. When finished, the teacher will ask the students for their feedback on the comic and clarify any words/sentences that students struggled to understand. Following this, the two activities (activity one being mandatory and activity two optional) associated with the respective comic will take place, with the teacher facilitating these. Once discussed and completed, the session will come to an end.

Statistical analyses

The full prospective Statistical Analysis Plan is summarised. Analyses will be conducted on an Intention-to-Treat (ITT) basis. Additional per protocol (PP) analyses will be performed. The per protocol analysis set will comprise those who provide outcome data and pass attention control checks requiring >= 80% of all attention control questions to be correctly answered. Missing data sensitivity analyses will be performed on both the ITT analysis set and the PP analysis set.

The primary outcome variable is the BESAA. The analysis plan for the secondary outcomes of the EDE-Q, Internalisation-General, BILD-Q, PANAS-C and RSES, and the exploratory outcome of endorsement of traditional gender norms will be the same as the BESAA. A linear mixed model will be used to examine the 2 by 2 by 2 factorial design (Randomized Arm [Control, Intervention], Phase [T2, T3], Gender [Male, Female]) using a hierarchically balanced model comprising all two-way interactions and two-way interactions with the baseline mean adjusted covariate. The model will additionally include school as a random factor, and a sensitivity analysis relating to the inclusion-exclusion of this effect will be conducted. Underpinning model assumptions will be examined. ANCOVA with mean adjusted baseline measure as covariate will be used to compare randomized arms at each of T2 and T3. The homogeneity of regression lines assumption will be assessed. In addition, separate sub-group analyses for boys and girls will be performed. Cohen's d and partial eta squared will be used to quantify standardised effect size, along with unadjusted means and 95% confidence intervals. Percentages reporting positive change, no change, and a poorer outcome, along with 95% confidence intervals will be reported. This study has multiple outcome measures (MOMs) at multiple time points. To limit serendipitous conclusions from MOMs, we will additionally report unadjusted p-values of the secondary outcomes at each of T2 and T3 along with results after controlling the False Discovery Rate (Benjamini & Hochberg, FDR using 0.2) and commit to reflecting this in the conclusions.

Exploratory analyses Exploratory outcome measures of skin colour dissatisfaction, body hair dissatisfaction, and appearance-based teasing, are single ordinal exploratory outcomes and will be compared between randomized groups at each of T2 and T3 using an ordinal logistic link controlling for baseline measures. Gender sub-group analyses will also be conducted.

Additionally, mediation analysis will be used to investigate whether interventional changes in Body Esteem between T1 and T3, and Body Esteem at T3, are mediated by changes in internalisation of appearance ideals between T1 and T2, and whether mediation is gender dependent.

EXTRA ANALYSES: Exploratory visual-based outcome measures of body size satisfaction and skin colour satisfaction are single ordinal exploratory outcomes and will be compared between randomized groups at each of T2 and T3 using an ordinal logistic link controlling for baseline measures. Gender sub-group analyses will also be conducted.

ELIGIBILITY:
Inclusion criteria for schools:

* Co-educational
* Located in semi-rural areas of Rajasthan
* Hindi-medium (i.e., Hindi should be the main medium of instruction)
* Include Classes 6-8 (students aged 11 to 14 years).

Exclusion criteria for schools:

* Single gender schools
* Located in urban areas of Rajasthan
* English medium
* Does not include Classes 6-8 (students aged 11 to 14 years).

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2631 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Body esteem: Validated Hindi language version of the Body Esteem Scale for adolescents & adults: Appearance and Weight subscales (Mendelson, Mendelson & White, 2001). | Baseline, post-intervention (4-weeks post baseline), 12-weeks follow-up
  Assessment of body esteem using the Appearance and Weight subscales from the Body Esteem Scale for adolescents & adults, 5-point Likert-type scale. Once the appropriate items are reverse coded, scores on all items are averaged; with lower scores indicating lower body esteem. This measure is currently undergoing validation among Indian adolescents and in Hindi language.

SECONDARY OUTCOMES:
Eating pathology: Validated Hindi language version of the Eating Disorder Examination Questionnaire (Fairburn & Wilson, 1993) | Baseline, post-intervention (4-weeks post baseline), 12-weeks follow-up
  Assessment of eating disorder pathology using the Eating Disorder Examination Questionnaire, 22 items, 7-point Likert-type scale. Scores on all items are averaged; with higher scores indicating greater eating pathology. This measure is currently undergoing validation among Indian adolescents and in Hindi language.
Internalisation of appearance ideals: Validated Hindi language version of the Sociocultural Attitudes Towards Appearance Questionnaire-3 (SATAQ-3): Internalisation-General subscale (Thompson et al., 2004) | Baseline, post-intervention (4-weeks post baseline), 12-weeks follow-up
  Assessment of internalisation of appearance ideals using the Internalisation-General subscale from the Sociocultural Attitudes Towards Appearance Questionnaire-3 (SATAQ-3):9 items, mean score range 1-5. Scores are averaged, with higher scores indicating higher internalisation. This measure is currently undergoing validation among Indian adolescents and in Hindi language.
Life disengagement due to body image concerns: Validated Hindi language version of the Body Image Life Disengagement Questionnaire (Atkinson & Diedrichs, 2021) | Baseline, post-intervention (4-weeks post baseline), 12-weeks follow-up
  Assessment of the extent to which worries or feeling bad about one's appearance has stopped the individual or is likely to stop them from engaging in life activities (e.g., going to a social event, doing physical activity, giving an opinion, going to school), 10 items, mean score range 1-4. Scores on all items are averaged; with higher scores indicating greater avoidance of activities due to appearance concerns.This measure is currently undergoing validation among Indian adolescents and in Hindi language.
Mood: Validated Hindi language version of the Positive and Negative Affect Scale - Children (Laurent et al., 1999) | Baseline, post-intervention (4-weeks post baseline), 12-weeks follow-up
  Assessment of both positive and negative mood using the Positive and Negative Affect Schedule - Children, 10 items, mean score range 1-5. Scores on the five items for the Positive Affect and Negative Affect subscales are averaged; with higher scores indicating greater negative affect and positive affect. This measure is currently undergoing validation among Indian adolescents and in Hindi language.
Self-esteem: Validated Hindi language version of the Rosenberg Self-Esteem Scale (Rosenberg, 1965) | Baseline, post-intervention (4-weeks post baseline), 12-weeks follow-up
  Assessment of self-esteem using the Short-Form Rosenberg Self-Esteem scale, 10 items, mean score range 1-4. Scores are averaged, with higher scores indicating greater self-esteem. This measure is currently undergoing validation among Indian adolescents and in Hindi language.

OTHER OUTCOMES:
Skin colour dissatisfaction: Purpose-built single-item measure developed for the study | Baseline, post-intervention (4-weeks post baseline), 12-weeks follow-up
  Assessment of skin colour dissatisfaction using a single-item measure ('How satisfied or dissatisfied are you with the colour of your skin?'), score range 1-5. This item will be in Hindi.
Body hair dissatisfaction: Purpose-built single-item measure developed for the study. | Baseline, post-intervention (4-weeks post baseline), 12-weeks follow-up
  Assessment of body hair dissatisfaction using a single-item measure ('How satisfied or dissatisfied are you with the amount of hair on your body?'), score range 1-5. This item will be in Hindi.
Appearance-based teasing: Single-item measure adapted from a previous body image intervention evaluation (Diedrichs et al, 2012). | Baseline, post-intervention (4-weeks post baseline), 12-weeks follow-up
  Assessment of appearance-based teasing using an item adapted from a previous body image intervention evaluation ('How often have you been teased about the way you look?'), score range 1-5. This item will be in Hindi.
Endorsement of traditional gender roles: A 10-item purpose built scale developed for the study and based on previous scales (Mills et al., 2012; Pulerwitz & Barker, 2008; Zeyneloglu & Terzioglu, 2011). | Baseline, post-intervention (4-weeks post baseline), 12-weeks follow-up
  Assessment of endorsement of traditional gender roles using a purpose-built measure based on previous scales. 10 items, mean score range 1-5. Scores are averaged, with higher scores indicating greater endorsement of traditional gender roles. This measure will be in Hindi.
ADDITIONAL: Body size satisfaction: Child Figure Rating Scale (Tiggemann & Wilson-Barrett, 1998) | Baseline, post-intervention (4-weeks post baseline), 12-weeks follow-up
  Visual-based assessment of body shape satisfaction, using discrepancy score between "ideal" and "perceived" figure (9 figures of varying body size). This measure will be in Hindi.
ADDITIONAL: Skin colour satisfaction: Purpose-built single-item measure developed for the study. | Baseline, post-intervention (4-weeks post baseline), 12-weeks follow-up
  Visual-based assessment of body shape satisfaction, using discrepancy score between "ideal" and "perceived" skin shade (9 varying skin shades from darker to lighter).This measure will be in Hindi.

CONTACTS AND LOCATIONS:
Overall Officials: Phillippa C Diedrichs, PhD, Principal Investigator — University of the West of England
Locations (1):
- Centre for Appearance Research, University of the West of England, Bristol, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Garbett KM, Lewis-Smith H, Chaudhry A, Shroff H, Dhillon M, White P, Diedrichs PC. Acceptability and preliminary efficacy of a school-based body image intervention in urban India: A pilot randomised controlled trial. Body Image. 2021 Jun;37:282-290. doi: 10.1016/j.bodyim.2021.02.011. Epub 2021 Apr 1. PMID 33813345
- [Result] Diedrichs PC, Atkinson MJ, Garbett KM, Leckie G. Evaluating the "Dove Confident Me" Five-Session Body Image Intervention Delivered by Teachers in Schools: A Cluster Randomized Controlled Effectiveness Trial. J Adolesc Health. 2021 Feb;68(2):331-341. doi: 10.1016/j.jadohealth.2020.10.001. Epub 2020 Nov 24. PMID 33243723
- [Derived] Lewis-Smith H, Ahuja L, Hasan F, Gentili C, White P, Diedrichs PC. A comic-based body image intervention for adolescents in semi-rural Indian schools: A randomised controlled trial. Int J Clin Health Psychol. 2025 Jan-Mar;25(1):100546. doi: 10.1016/j.ijchp.2025.100546. Epub 2025 Jan 26. PMID 39911164
- [Derived] Ahuja L, Hasan F, Diedrichs PC, Lewis-Smith H. Comics as a body image intervention among adolescents in Indian Hindi medium schools: insights from an acceptability study. Glob Ment Health (Camb). 2022 Sep 29;9:460-469. doi: 10.1017/gmh.2022.50. eCollection 2022. PMID 36618749

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-06-09): https://cdn.clinicaltrials.gov/large-docs/55/NCT04317755/SAP_000.pdf